CLINICAL TRIAL: NCT01007448
Title: Phase IV Randomized Study of Two Dose Levels of Targretin® Capsules in Subjects With Refractory Cutaneous T-Cell Lymphoma
Brief Title: Study Evaluating Two Dose Levels of Targretin Capsules in Participants With Refractory Cutaneous T-Cell Lymphoma (CTCL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7273-G000-401
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Refractory Cutaneous T-cell Lymphoma
Keywords: CTCL; bexarotene; Targretin; Refractory Cutaneous T-cell Lymphoma; cutaneous T-cell Lymphoma; MF; Mycoses fungoides
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides | interventions — Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bexarotene 150 milligrams (mg)/square meter (m^2)/day (Experimental): Participants will receive bexarotene 150 mg/m^2/day once daily for 24 weeks.
  Interventions: Drug: Bexarotene
- Bexarotene 300 mg/m^2/day (Experimental): Participants will receive bexarotene 300 mg/m^2/day once daily for 24 weeks.
  Interventions: Drug: Bexarotene

INTERVENTIONS:
Drug: Bexarotene — Soft gelatin capsules to be taken orally with at least 6 ounces of water or other fluid either with or immediately following the evening meal (a moderate or full meal) or a nutritionally defined liquid food.
  Other Names: Targretin®

SUMMARY:
This is a multicenter, randomized, open-label, Phase IV study to assess the efficacy, tolerability, and safety of 2 initial dose levels of bexarotene capsules in participants with refractory CTCL.

ELIGIBILITY:
Inclusion Criteria:

1. A CTCL without central nervous system (CNS) involvement, confirmed by biopsy to be histologically consistent with CTCL diagnosis by a dermatopathologist.
2. Refractory to at least 1 systemic therapy for CTCL. (Refractory is defined as resistance to therapy due either to lack of response of at least 50% improvement or progression of disease while still on therapy after an initial response.)
3. Systemic therapy for CTCL is indicated.
4. A Karnofsky performance score ≥60%.
5. Age ≥18 years.
6. Females of childbearing potential must have a negative serum beta human chorionic gonadotropin (ß-hCG) with a sensitivity of at least 50 milli-international units/liter (mIU/L) within 7 days prior to the initiation of treatment. Females of childbearing potential must have used simultaneously two highly effective methods of contraception (strongly recommended that 1 of the 2 forms of contraception be non-hormonal such as condom plus spermicide, condom plus diaphragm with spermicide, or have a vasectomized partner) or use an intrauterine device or must have been sexually abstinent for at least four weeks prior to or at least 1 menstrual cycle prior to (whichever is longer) the negative pregnancy test through entry in the study. Sexual abstinence or effective contraception must be used for at least 1 month prior to the initiation of therapy, during therapy, and for at least 1 month following discontinuation of therapy. Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
7. Male participants with female partners of childbearing potential must agree to sexual abstinence or to practice 2 reliable forms of effective contraception used simultaneously (strongly recommended that 1 of the 2 forms of contraception be non-hormonal such as condom plus spermicide, condom plus diaphragm with spermicide, or partner with tubal ligation) or partner may use an intrauterine device, during the entire period of bexarotene capsule treatment and for at least 1 month after treatment is discontinued. Male participants with female sexual partners who are pregnant, possibly pregnant or who could become pregnant during the study must agree to use condoms during sexual intercourse during the entire period of bexarotene capsule treatment and for at least 1 month after the last dose of bexarotene capsules.
8. Must be willing and able to give informed consent and complete and understand, either oral or written, study procedures and assessments.
9. Participant must be suitable for participation in the study in the Investigator's opinion.
10. Fasting serum triglyceride within normal limits (<150 mg/deciliter [dL]) prior to study entry.
11. Adequate renal function as evidenced by serum creatinine ≤2.0 mg/dL or calculated creatinine clearance ≥40 milliliters (mL)/minute (min) as per the Cockroft and Gault formula.
12. Adequate hepatic function that is characterized by aspartate aminotransferase (SGOT [AST]), alanine aminotransferase (SGPT [ALT]), or serum bilirubin <2.5 times the upper limit of normal.
13. Adequate bone marrow function as evidenced by hemoglobin ≥8 grams (g)/dL, absolute neutrophil count (ANC) ≥1,000/milliliters cubed (mm^3), and platelets ≥50,000/mm^3.

Exclusion Criteria

1. Cutaneous T-cell lymphoma involving the central nervous system.
2. Participants with known Human Immunodeficiency Virus (HIV) infection and active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection (HBV/HCV or HIV testing is not required for the purpose of this study).
3. Participation in any other investigational drug study within 30 days of entry in this study.
4. Within 5 years after the onset of menopause.
5. Received systemic corticosteroids within 6 months of entry in the study.
6. Known hypersensitivity to bexarotene or other component of bexarotene capsules.
7. Pregnancy, intent to become pregnant, or breast-feeding.
8. Received gemfibrozil within 1 day of starting the study.
9. Prior therapy for the treatment of CTCL:

   1. Psoralens and ultraviolet A light (PUVA) or ultraviolet B light (UVB) therapy within 3 weeks of study entry.
   2. Electron beam radiation therapy (EBT) or photopheresis within 3 weeks of study entry.
   3. Topical retinoids, nitrogen mustard, carmustine (BCNU), imiquimod, or other antipruritic medication within 2 weeks of study entry.

      If antipruritic medication cannot be avoided, antihistamine or antipruritic agents must be administered using a stable dose regimen for at least 1 week prior to initiation of study drug treatment and throughout the study, unless it is determined that a discontinuation or reduction in dose is indicated. Prior to the enrollment of any participant who will be taking systemic or dermatologically-applied antihistamine or anti-pruritic agent, the investigator must contact Eisai to discuss the need for such agent. Mineral oil, baby oil, and simple moisturizing lotions may be used as emollients. Low- to mid- potency topical corticosteroids are allowed only for participants with erythroderma (Stage III/IV CTCL) using a stable dose regimen for at least 4 weeks prior to study entry. High potency topical corticosteroids and tar baths are NOT permitted.

      NOTE: Prior to the enrollment of any participant who will be taking systemic or dermatologically-applied antihistamine or anti-pruritic agent, the Investigator must contact the Sponsor to discuss the need for such agent.
   4. Anticancer therapy of any kind (for example, methotrexate, cyclophosphamide, vorinostat, romidepsin, and interferon) within 30 days of entry to the study. Participant must recover from all signs of toxicity prior to entry in the study.
   5. Oral retinoid therapy for any indication within 3 months of study entry.
   6. Systemic therapy with Vitamin A in doses of greater than 15,000 International Units (IU) (5,000 microgram [mcg]) per day (equivalent to approximately 3 times Recommended Daily Allowance [RDA]) within 30 days of entry in this study.
10. Systemic antibiotic therapy within 2 weeks of entry in the study. (Participants with infections requiring antibiotics or likely to require antibiotics should be appropriately treated with a course of antibiotics terminating at least two weeks prior to entry, or if indicated, a chronic suppressive or prophylactic dose of antibiotics stabilized at least 2 weeks prior to entry. Participants who require initiation of or changes in antibiotic therapy during the study will not be considered a violation of the study protocol).
11. History of pancreatitis or significant risk factors for developing pancreatitis (for example, prior pancreatitis, uncontrolled hyperlipidemia, excessive alcohol consumption, uncontrolled diabetes mellitus, biliary tract disease, and medications known to increase triglyceride levels or to be associated with pancreatic toxicity).
12. Unwillingness or inability to minimize exposure to sunlight and artificial ultraviolet light while receiving bexarotene capsules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-01-06 (Actual); Primary Completion 2014-02-20 (Actual); Study Completion 2014-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Kaur, MD, Study Director — Valeant Pharmaceutical NA
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Florida Academic Dermatology Centers, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - Tulane, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University Health, Winston-Salem, North Carolina
  - University Hospitals-Case Medical Center, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute At the University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1 ratio to bexarotene 150 milligrams (mg)/square meter (m^2)/day or 300 mg/m^2/day.
Groups:
- Bexarotene 150 mg/m^2/Day: Participants received bexarotene 150 mg/m^2/day once daily for 24 weeks.
- Bexarotene 300 mg/m^2/Day: Participants received bexarotene 300 mg/m^2/day once daily for 24 weeks.
Period: Overall Study
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Started | 30 | 29
Full Analysis Population (Received at Least 1 Dose of Study Drug) | 30 | 29
Safety Population (Received at Least 1 Dose of Study Drug and had at least 1 safety assessment after treatment.) | 30 | 29
Completed | 20 | 20
Not Completed | 10 | 9
Not completed — Continuing Prohibited Systemic Drugs | 1 | 0
Not completed — Staph Skin Infection Flare | 1 | 0
Not completed — Participant Leaving the Country | 1 | 0
Not completed — Participant Given Prohibited Medication | 1 | 0
Not completed — Progressive Disease | 1 | 2
Not completed — Lack of Efficacy | 2 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 1 | 4

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug (Full Analysis Population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (14.80) | 61.0 (13.94) | 60.6 (14.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tumor Response (Complete Response [CR], Clinical Complete Response [CCR], and Partial Response [PR]) in up to 5 Index Lesions as Determined by Investigator's Composite Assessment (CA) of Index Lesion Disease Severity
Description: Index lesion symptoms/grade include: erythema=0 (no evidence)-8 (very severe); scaling=0 (no evidence)-8 (very severe); plaque elevation=0 (no evidence)-8 (extreme elevation); hypopigmentation/hyperpigmentation=0 (no evidence of change)-8 (very severe change); area of involvement=0 (0 centimeters [cm]^2)-18 (>300 cm^2). CA generated by sum of grades of signs/symptoms for each index lesion. Index lesion CA grade at baseline was divided into CA grade at each subsequent study visit to determine participant's response to treatment. Ratio of CA <1.0=improvement in disease; ratio >1.0=worsening of disease. Tumor response as determined by CA=percentage of participants achieving CR (CA ratio=0, no clinically abnormal lymph nodes, and absence of histologic signs of CTCL); CCR (CA ratio=0 and no clinically abnormal lymph nodes); and PR (CA ratio=≤0.5, <25% increase in number/aggregate area of abnormal lymph nodes/tumors, and no new abnormal lymph nodes in documented area of absence of disease).
Time Frame: Baseline up to Week 24
Population: Participants who received at least 1 dose of study drug (Full Analysis Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Number analyzed (Participants) | 30 | 29
Participants
  CR | 0 | 0
  CCR | 2 | 3
  PR | 5 | 7

2. Primary Outcome: Number of Participants With Tumor Response of CR, CCR, PR, SD, and PD as Determined by Physician's Global Assessment (PGA) of Clinical Condition
Description: The PGA was an assessment of the overall extent of improvement/worsening from Baseline of the participant's overall disease compared with the condition every 4 weeks thereafter during treatment. CR=PGA grade of 0 (completely clear of disease since Baseline) and absence of histologic signs of CTCL. CCR=PGA grade of 0. PR=PGA grade of 1 (almost clear [≥90%-<100%] of disease since Baseline), 2 (marked improvement [≥75%-<90%] of disease since Baseline), 3 (moderate improvement [≥50%-<70%] of disease since Baseline). Stable Disease (SD)=PGA grade of 4 (slight improvement [<25%-<50%] of disease since Baseline) or 5 (no change in disease [+/-<25% change since Baseline]). Progressive Disease (PD)=PGA grade of 6 (worse disease [≥25%] than at baseline). If visceral disease or an abnormal lymph node was located in a documented area of absence of disease, then PD would be reported for the participant.
Time Frame: Baseline up to Week 24
Population: Participants who received at least 1 dose of study drug (Full Analysis Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Number analyzed (Participants) | 30 | 29
Participants
  CR | 0 | 0
  CCR | 1 | 3
  PR | 5 | 8
  SD | 23 | 16
  PD | 0 | 0
  Unknown | 1 | 2

3. Primary Outcome: Number of Participants With Tumor Response of CR, CCR, PR, SD, and PD as Determined Percent Body Surface Area (BSA) Involvement
Description: To determine BSA involvement, the area of the participant's palm was defined as 1% of the participant's BSA. The extent of involvement of disease was determined as multiples of the participant's palm area and expressed as a percentage of the participant's total BSA at Baseline (Day 1) and every 4 weeks thereafter during treatment. CR=percent BSA 0% and documented absence of histologic signs of CTCL. CCR=Percent BSA 0%. PR=a decrease from Baseline in percent BSA of at least 50%. SD=none of the response classifications (that is, CR, CCR, PR, or PD) accurately describe the disease status. PD=an increase from Baseline in percent BSA of at least 25%.
Time Frame: Baseline up to Week 24
Population: Participants who received at least 1 dose of study drug (Full Analysis Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Number analyzed (Participants) | 30 | 29
Participants
  CR | 1 | 2
  CCR | 0 | 1
  PR | 6 | 7
  SD | 22 | 17
  PD | 0 | 0
  Unknown | 1 | 2

4. Secondary Outcome: Duration of Tumor Response (CR, CCR, or PR) as Determined by Investigator's CA of Index Lesion Disease Severity
Description: Defined as time interval from onset of response to time participant relapses or last date of data collected with an assessment of participant still meeting response criteria. Index lesion symptoms/grade: erythema/scaling=0 (no evidence)-8 (very severe); plaque elevation=0 (no evidence)-8 (extreme elevation); hypopigmentation/hyperpigmentation=0 (no evidence)-8 (very severe change); area of involvement=0 (0 cm^2)-18 (>300 cm^2). CA: sum of signs/symptoms grades for index lesion. Index lesion CA grade at baseline divided into CA grade at study visit to determine treatment response. CA Ratio <1.0=improvement and >1.0=worsening of disease. Tumor response=percentage of participants with CR (CA ratio=0, no clinically abnormal lymph nodes, absence of CTCL histologic signs); CCR (CA ratio=0; no clinically abnormal lymph nodes); PR (CA ratio=≤0.5, <25% increase in number/aggregate area of abnormal lymph nodes/tumors, no new abnormal lymph nodes in documented area of absence of disease).
Time Frame: Baseline up to Week 24
Population: Participants who received at least 1 dose of study drug (Full Analysis Population) and with the best overall response of evaluable CR, CCR, and PR data for CA of index lesion disease severity.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Number analyzed (Participants) | 7 | 10
days | 65.9 (41.86) | 83.7 (36.50)

5. Secondary Outcome: Duration of Tumor Response (CR, CCR, or PR) as Determined by PGA of Clinical Condition
Description: Defined as time interval from onset of response to time participant relapses or last date of data collected with an assessment of participant still meeting response criteria. PGA was an assessment of the overall extent of improvement/worsening from Baseline of the participant's overall disease compared with the condition every 4 weeks thereafter during treatment. CR=PGA grade of 0 (completely clear of disease since Baseline) and absence of histologic signs of CTCL. CCR=PGA grade of 0. PR=PGA grade of 1 (almost clear [≥90%-<100%] of disease since Baseline), 2 (marked improvement [≥75%-<90%] of disease since Baseline), 3 (moderate improvement [≥50%-<70%] of disease since Baseline).
Time Frame: Baseline up to Week 24
Population: Participants who received at least 1 dose of study drug (Full Analysis Population) and with the best overall response of evaluable CR, CCR, and PR data for PGA of clinical condition.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Number analyzed (Participants) | 6 | 11
days | 111.5 (34.61) | 69.4 (38.93)

6. Secondary Outcome: Duration of Tumor Response (CR, CCR, or PR) as Determined by Percent BSA Involvement
Description: Defined as time interval from onset of response to time participant relapses or last date of data collected with an assessment of participant still meeting response criteria. To determine BSA, the area of the participant's palm was defined as 1% of the participant's BSA. The extent of involvement of disease was determined as multiples of the participant's palm area and expressed as a percentage of the participant's total BSA at Baseline (Day 1) and every 4 weeks thereafter during treatment. CR=percent BSA 0% and documented absence of histologic signs of CTCL. CCR=Percent BSA 0%. PR=a decrease from Baseline in percent BSA of at least 50%.
Time Frame: Baseline up to Week 24
Population: Participants who received at least 1 dose of study drug (Full Analysis Population) and with the best overall response of evaluable CR, CCR, and PR data for percent of BSA involvement.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Number analyzed (Participants) | 7 | 10
days | 99.4 (41.69) | 54.1 (42.18)

7. Secondary Outcome: Time to Tumor Response (CR, CCR, or PR) as Determined by CA of Index Lesion Disease Severity
Description: Defined as time interval from first day of bexarotene treatment to time of first observation when participant met the criteria of CR, CCR, or PR. Index lesion symptoms/grade: erythema/scaling=0 (no evidence)-8 (very severe); plaque elevation=0 (no evidence)-8 (extreme elevation); hypopigmentation/hyperpigmentation=0 (no evidence)-8 (very severe change); and area of involvement=0 (0 cm^2)-18 (>300 cm^2). CA: sum of signs/symptoms grades for index lesion. Index lesion CA grade at baseline divided into CA grade at study visit to determine treatment response. CA Ratio <1.0=improvement and >1.0=worsening of disease. Tumor response=percentage of participants with CR (CA ratio=0, no clinically abnormal lymph nodes, and absence of CTCL histologic signs); CCR (CA ratio=0 and no clinically abnormal lymph nodes); and PR (CA ratio=≤0.5, <25% increase in number/aggregate area of abnormal lymph nodes/tumors, and no new abnormal lymph nodes in documented area of absence of disease).
Time Frame: Baseline up to Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Number analyzed (Participants) | 7 | 10
days | 99.9 (39.14) | 91.6 (37.20)

8. Secondary Outcome: Time to Tumor Response (CR, CCR, or PR) as Determined by PGA of Clinical Condition
Description: Defined as time interval from first day of bexarotene treatment to time of first observation when participant met the criteria of CR, CCR, or PR. PGA was an assessment of the overall extent of improvement/worsening from Baseline of the participant's overall disease compared with the condition every 4 weeks thereafter during treatment. CR=PGA grade of 0 (completely clear of disease since Baseline) and absence of histologic signs of CTCL. CCR=PGA grade of 0. PR=PGA grade of 1 (almost clear [≥90%-<100%] of disease since Baseline), 2 (marked improvement [≥75%-<90%] of disease since Baseline), 3 (moderate improvement [≥50%-<70%] of disease since Baseline).
Time Frame: Baseline up to Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Number analyzed (Participants) | 6 | 11
days | 53.5 (23.32) | 103.5 (41.34)

9. Secondary Outcome: Time to Tumor Response (CR, CCR, or PR) as Determined by Percent BSA Involvement
Description: Defined as time interval from first day of bexarotene treatment to time of first observation when participant met the criteria of CR, CCR, or PR. To determine BSA, the area of the participant's palm was defined as 1% of the participant's BSA. The extent of involvement of disease was determined as multiples of the participant's palm area and expressed as a percentage of the participant's total BSA at Baseline (Day 1) and every 4 weeks thereafter during treatment. CR=percent BSA 0% and documented absence of histologic signs of CTCL. CCR=Percent BSA 0%. PR=a decrease from Baseline in percent BSA of at least 50%.
Time Frame: Baseline up to Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Number analyzed (Participants) | 7 | 10
days | 66.1 (36.97) | 117.0 (41.90)

10. Secondary Outcome: Time to Tumor Progression as Determined by CA of Index Lesion Disease Severity
Description: Defined as time interval from first day of bexarotene treatment to time of first observation when participant met criteria for PD. Index lesion symptoms/grade: erythema/scaling=0 (no evidence)-8 (very severe); plaque elevation=0 (no evidence)-8 (extreme elevation); hypopigmentation/hyperpigmentation=0 (no evidence)-8 (very severe change); and area of involvement=0 (0 cm^2)-18 (>300 cm^2). CA: sum of signs/symptoms grades for index lesion. Index lesion CA grade at baseline divided into CA grade at study visit to determine treatment response. CA Ratio <1.0=improvement and >1.0=worsening of disease. Criteria for PD requires at least 1 component of the following: CA ratio=≥1.25, ≥25% increase in number/aggregate area of abnormal lymph nodes/tumors, or no new abnormal lymph nodes in documented area of absence of disease.
Time Frame: Baseline up to Week 24
Population: Participants who received at least 1 dose of study drug (Full Analysis Population) and with evaluable PD data for CA of index lesion disease severity.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Number analyzed (Participants) | 1 | 2
days | 203.0 (NA) — NA=Not available. Standard deviation cannot be calculated with an N of 1. | 77.5 (58.69)

11. Secondary Outcome: Time to Tumor Progression as Determined by PGA of Clinical Condition
Description: Defined as time interval from first day of bexarotene treatment to time of first observation when participant met criteria for PD. PGA was an assessment of the overall extent of improvement/worsening from Baseline of the participant's overall disease compared with the condition every 4 weeks thereafter during treatment. PD=PGA grade of 6 (worse disease [≥25%] than at baseline). If visceral disease or an abnormal lymph node was located in a documented area of absence of disease, then PD would be reported for the participant.
Time Frame: Baseline up to Week 24
Population: Participants who received at least 1 dose of study drug (Full Analysis Population) and with progression.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Number analyzed (Participants) | 0 | 2
days |  | 115.5 (4.95)

12. Secondary Outcome: Time to Tumor Progression as Determined by Percent BSA Involvement
Description: Defined as time interval from first day of bexarotene treatment to time of first observation when participant met criteria for PD. To determine BSA involvement, the area of the participant's palm was defined as 1% of the participant's BSA. The extent of involvement of disease was determined as multiples of the participant's palm area and expressed as a percentage of the participant's total BSA at Baseline (Day 1) and every 4 weeks thereafter during treatment. PD=an increase from Baseline in percent BSA of at least 25%.
Time Frame: Baseline up to Week 24
Population: Participants who received at least 1 dose of study drug (Full Analysis Population) and with progression.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Number analyzed (Participants) | 2 | 2
days | 86.0 (1.41) | 88.0 (43.84)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 28
Description: Received at Least 1 Dose of Study Drug and had at least 1 safety assessment after treatment (Safety Population).
Arm/Group | Bexarotene 150 mg/m^2/Day | Bexarotene 300 mg/m^2/Day
Serious Adverse Events (participants affected / at risk) | 11/30 | 13/29
Other Adverse Events (participants affected / at risk) | 21/30 | 21/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bexarotene 150 mg/m^2/Day (N=30) | Bexarotene 300 mg/m^2/Day (N=29)
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 9
Renal failure (Renal and urinary disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bexarotene 150 mg/m^2/Day (N=30) | Bexarotene 300 mg/m^2/Day (N=29)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 17 | 14
Hypothyroidism (Endocrine disorders) | 12 | 15
Headache (Nervous system disorders) | 7 | 9
Hypercholesterolemia (Metabolism and nutrition disorders) | 7 | 7
Skin exfoliation (Skin and subcutaneous tissue disorders) | 5 | 5
Neutropenia (Blood and lymphatic system disorders) | 2 | 5
Blood triglycerides increased (Investigations) | 3 | 4
Thyroxine free decreased (Investigations) | 4 | 4
Alanine aminotransferase increased (Investigations) | 3 | 4
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 3
Oedema peripheral (General disorders) | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Bacterial test positive (Investigations) | 4 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 3
Fatigue (General disorders) | 2 | 2
Urinary tract infection (Infections and infestations) | 3 | 1
White blood cell count decreased (Investigations) | 2 | 2
Hypertension (Vascular disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 2
Neutrophil count decreased (Investigations) | 3 | 0
Sinusitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Lethargy (Nervous system disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Pnemonia (Infections and infestations) | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.